CLINICAL TRIAL: NCT06844539
Title: Targeting Beta-cell Function to Achieve Remission of Type 2 Diabetes (REACTIVATE). An Open-label, Single-centre, Randomised, Parallel Study to Assess the Efficacy, Safety and Utility of Fully Closed-loop Insulin Delivery in Achieving Remission of Diabetes Compared to Standard Therapy With a Glucose Sensor in Adults With Recent Onset Type 2 Diabetes
Brief Title: taRgeting bEtA-Cell Function To achIeVe Remission of Type 2 diAbeTEs
Acronym: REACTIVATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Charlotte Boughton, Clinical Research Associate, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REACTIVATE 346139
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
Keywords: Remission; closed-loop
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fully automated insulin delivery (Experimental): Fully automated insulin delivery with CamAPS HX, Freestyle Libre 3 Sensor and Ypsopump insulin pump for 12 weeks
  Interventions: Device: Fully automated insulin delivery with CamAPS HX
- Standard therapy with a glucose sensor (Active Comparator): Standard diabetes therapy with a glucose sensor for 12 weeks
  Interventions: Device: Standard diabetes therapy with a glucose sensor

INTERVENTIONS:
Device: Fully automated insulin delivery with CamAPS HX — Fully automated insulin delivery with CamAPS HX app, Libre 3 glucose sensor and Ypsopump insulin pump.
  Arms: Fully automated insulin delivery
Device: Standard diabetes therapy with a glucose sensor — Standard diabetes therapy with a Freestyle Libre 3 glucose sensor
  Arms: Standard therapy with a glucose sensor

SUMMARY:
The main objective of the REACTIVATE study is to investigate whether a period of intensive insulin therapy using closed-loop technology, when combined with diet and lifestyle education, can restore beta-cell function and achieve remission of recent-onset type 2 diabetes.

This is a single-centre, open-label, randomised, parallel design study comparing up to 12 weeks of fully closed-loop insulin delivery to standard care with a glucose sensor in adults with recent-onset type 2 diabetes. The primary outcome is the number of participants achieving remission of diabetes at 52 weeks, defined as HbA1c below 48mmol/mol after 12 or more weeks off all diabetes medications.

Other key outcomes include area under the curve for C-peptide and glucose during mixed meal tolerance test, the proportion of time spent with glucose levels within and above the target glucose range and mean sensor glucose as recorded by glucose sensor at 52 weeks.

Safety evaluation comprises severe hypoglycaemic episodes, and other adverse and serious adverse events. Utility and human factors outcomes include glucose sensor and closed-loop usage, questionnaires and semi-structured interviews.

DETAILED DESCRIPTION:
This is a single-centre, open-label, randomised, parallel design study comparing up to 12 weeks of fully closed-loop insulin delivery to standard care with a glucose sensor in adults with recent-onset type 2 diabetes.

Recruitment will target up to 56 participants to allow for drop-outs. Participants will be recruited from outpatient clinics at Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, local GP surgeries, social media advertising or other established practices at the centre. Written informed consent will be obtained from all participants before any study related activities.

After obtaining informed consent, the baseline visit (including mixed meal tolerance test) and a 2-3 week run-in period, participants will be randomised to either 12 weeks use of fully closed-loop insulin delivery or 12 weeks during which they will apply their standard diabetes therapy with a glucose sensor. Participants in both groups will receive diet and lifestyle advice with specific focus on the impact of diet and lifestyle choices on glucose sensor readings and trends.

Following the 12 weeks intervention period (and repeat mixed meal tolerance test) all participants will continue with standard diabetes therapy for nine months of follow-up (and final mixed meal tolerance test). Diabetes therapies will be adjusted every 3 months based on HbA1c.

The study includes up to 5 visits and 6 telephone/email contacts. Visits 2 and 3 may be combined. All participants will continue to be seen by their clinical team at frequencies as appropriate in line with usual clinical practice. All study visits will be scheduled in addition to routine clinical visits and will be performed by the research team. Maximum time in the study is 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Type 2 diabetes diagnosed >6 months and ≤5 years ago
* Treatment with glucose lowering medication for at least 3 months
* HbA1c >48 mmol/mol on analysis from local laboratory or equivalent
* Willing to wear study devices and follow study instructions
* Capacity to consent to participate in the study

Exclusion Criteria:

* Type 1 diabetes
* Current use of insulin pump
* Current use of any closed-loop system
* Any physical/psychological disease or medication(s) likely to interfere with the conduct of the study and interpretation of the study results, as judged by study clinician
* Known or suspected allergy against insulin
* Pregnancy, planned pregnancy, or breast feeding
* Severe visual or hearing impairment
* Medically documented allergy towards the adhesive of plasters
* Serious skin diseases located at places of the body potentially used for localisation of the glucose sensor
* Drug or alcohol misuse
* Group 2 driving licence holder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-04-24 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
The number of participants achieving remission of diabetes at 52 weeks | 52 weeks
  The between group difference in the number of participants achieving remission of diabetes at 52 weeks, defined as HbA1c <48mmol/mol after ≥12 weeks off all diabetes medications.

SECONDARY OUTCOMES:
Mixed meal tolerance test (MMTT) area under the curve for C-peptide | 12 weeks
  Mixed meal tolerance test (MMTT) area under the curve for C-peptide
Mixed meal tolerance test (MMTT) area under the curve for C-peptide | 52 weeks
  Mixed meal tolerance test (MMTT) area under the curve for C-peptide
Mixed meal tolerance test (MMTT) area under the curve for glucose | 12 weeks
  Mixed meal tolerance test (MMTT) area under the curve for glucose
Mixed meal tolerance test (MMTT) area under the curve for glucose | 52 weeks
  Mixed meal tolerance test (MMTT) area under the curve for glucose
Proportion of time spent in tight target glucose range (3.9 to 7.8mmol/l) | 12 weeks
  Proportion of time spent with sensor glucose in tight target glucose range (3.9 to 7.8mmol/l)
Proportion of time spent in tight target glucose range (3.9 to 7.8mmol/l) | 52 weeks
  Proportion of time spent with sensor glucose in tight target glucose range (3.9 to 7.8mmol/l)
Proportion of time spent in target glucose range (3.9 to 10.0mmol/l) | 12 weeks
  Proportion of time spent with sensor glucose in target glucose range (3.9 to 10.0mmol/l)
Proportion of time spent intarget glucose range (3.9 to 10.0mmol/l) | 52 weeks
  Proportion of time spent with sensor glucose in target glucose range (3.9 to 10.0mmol/l)
Proportion of time spent below target glucose range (<3.9mmol/l) | 12 weeks
  Proportion of time spent below target glucose range (<3.9mmol/l)
Proportion of time spent below target glucose range (<3.9mmol/l) | 52 weeks
  Proportion of time spent below target glucose range (<3.9mmol/l)
Proportion of time spent above target glucose range (>10.0mmol/l) | 12 weeks
  Proportion of time spent above target glucose range (>10.0mmol/l)
Proportion of time spent above target glucose range (>10.0mmol/l) | 52 weeks
  Proportion of time spent above target glucose range (>10.0mmol/l)
Mean sensor glucose | 12 weeks
  Mean sensor glucose (mmol/l)
Mean sensor glucose | 52 weeks
  Mean sensor glucose (mmol/l)
Glycated haemoglobin | 12 weeks
  HbA1c (mmol/mol)
Glycated haemoglobin | 52 weeks
  HbA1c (mmol/mol)
Blood pressure | 12 weeks
  Blood pressure (mmHg)
Blood pressure | 52 weeks
  Blood pressure (mmHg)
Body weight | 12 weeks
  Body weight (kg)
Body weight | 52 weeks
  Body weight (kg)
Number of diabetes medications | 52 weeks
  Number of diabetes medications

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte K Boughton, Principal Investigator — University of Cambridge
Locations (1):
- Addenbrooke's Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to cb2000@cam.ac.uk and may be submitted up to 36 months following article publication. To gain access, data requestors will need to sign a data access agreement.
  Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to cb2000@cam.ac.uk and may be submitted up to 36 months following article publication.
Access Criteria: Study protocol, statistical analysis plan and fully anonymised individual participant data that underlie the results reported in the manuscript will be available 6 months following publication and ending 36 months following manuscript publication to investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose, to achieve aims in the approved proposal. Proposals should be directed to cb2000@cam.ac.uk and may be submitted up to 36 months following article publication.